CLINICAL TRIAL: NCT04321278
Title: Evaluation of the Safety and Clinical Efficacy of Hydroxychloroquine Associated With Azithromycin in Patients With Pneumonia Caused by Infection by the SARS-CoV2 Virus - Coalition COVID-19 Brasil II - SEVERE - Patients
Brief Title: Safety and Efficacy of Hydroxychloroquine Associated With Azithromycin in SARS-CoV2 Virus (Coalition Covid-19 Brasil II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: EMS (Industry); Hospital do Coracao (Other); Hospital Sirio-Libanes (Other); Brazilian Research In Intensive Care Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30155020.5.1001.0071
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Infections; Pneumonia, Viral
Keywords: SARS-CoV2 virus; 2019-nCOV; COVID-19; hydroxychloroquine; azithromycin
MeSH Terms: conditions — Coronavirus Infections; Pneumonia, Viral; COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Intervention Model Description: 1. Intervention Group: Hydroxychloroquine + azithromycin. After randomization, Hydroxychloroquine [400mg 2x/day, 12/12h] + azithromycin [500mg 1x/day]) for 10 days. Standard treatment is according to the treatment protocol for 2019-nCoV infection.
  2. Active Control Group: Hydroxychloroquine. After randomization, Hydroxychloroquine [400mg 2x/day, 12/12h] for 10 days. Standard treatment is according to the treatment protocol for 2019-nCoV infection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine + azithromycin (Experimental): Hydroxychloroquine [400mg 2x/day, 12/12h] + azithromycin [500mg 1x/day]
  Interventions: Drug: Hydroxychloroquine + azithromycin
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine [400mg 2x/day, 12/12h]
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine + azithromycin — Intervention Group: Hydroxychloroquine + azithromycin. After randomization, Hydroxychloroquine [400mg 2x/day, 12/12h] + azithromycin [500mg 1x/day]) for 10 days. Standard treatment is according to the treatment protocol for 2019-nCoV infection.
  Other Names: HCQ+AZI
  Arms: Hydroxychloroquine + azithromycin
Drug: Hydroxychloroquine — Active Control Group: Hydroxychloroquine. After randomization, Hydroxychloroquine [400mg 2x/day, 12/12h] for 10 days. Standard treatment is according to the treatment protocol for 2019-nCoV infection.
  Other Names: HCQ
  Arms: Hydroxychloroquine

SUMMARY:
The Severe Acute Respiratory Syndrome COronaVirus 2 (SARS-CoV2) is a new and recognized infectious disease of the respiratory tract. Around 20% of those infected have severe pneumonia and currently there is no specific or effective therapy to treat this disease. Therapeutic options using malaria drugs chloroquine and hydroxychloroquine have shown promising results in vitro and in vivo test. But those efforts have not involved large, carefully-conducted controlled studies that would provide the global medical community the proof that these drugs work on a significant scale. In this way, the present study will evaluate the effectiveness and safety of the use of hydroxychloroquine combined with azithromycin compared to hydroxychloroquine monotherapy in patients hospitalized with pneumonia by SARS-CoV2 virus.

DETAILED DESCRIPTION:
The Severe Acute Respiratory Syndrome COronaVirus 2 (SARS-CoV2) is a new and recognized infectious disease of the respiratory tract that is now spreading to several countries in the world, including Brazil. Mortality rates after infection are higher in adults over 60 and with a history of comorbidities. The most serious patients need care in intensive care units (ICU). Most of the time they depend on mechanical ventilation support due to acute respiratory distress syndrome (ARDS). Infection rates are higher than the capacity for intensive care, which represents a serious problem in medical care. Around 20% of those infected have severe pneumonia and so far it does not have a specific therapy, or even, an effective clinical management. Therapeutic options using malaria drugs chloroquine and hydroxychloroquine have shown promising results in vitro and in vivo test. A recent, small, non-randomized study with hydroxychloroquine in 36 patients infected with SARS-Cov-2 proved to be promising in the ability to reset the viral load in 6 days after starting treatment. Thus, the present study will evaluate the effectiveness and safety of the use of hydroxychloroquine combined with azithromycin compared to hydroxychloroquine monotherapy in the clinical evolution by the ordinal scale of 6 points in adult patients hospitalized with pneumonia caused by infection by the SARS-CoV2 virus in Brazil.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged > 18 years;
2. Suspected or confirmed infection by SARS-CoV2;

Presenting with one of the following:

* Need for oxygen supplementation > 4 L/min, or
* Need for high-flow nasal canula, or
* Need for non-invasive ventilation, or
* Need for mechanical ventilation.

Exclusion Criteria:

1. Refusal to provide written informed consent (either the patient or a legal representative);
2. Hypersensitivity to any of the drugs used in the study (Azithromycin or Hydroxychloroquine);
3. Patients with more than 48 hours of prior study medication use;
4. Patients with onset of symptoms longer than 14 days;
5. Patients with long QT syndrome or severe ventricular arrhythmias, not protected by an implantable cardioverter defibrillators (ICD).;
6. QTc>= 480ms;
7. Do not resuscitate order or exclusive palliative care;
8. Patients with liver disease or cirrhosis or abnormal liver enzyme tests above three times the upper limit values (alanine aminotransferase -ALT and aspartate aminotransferase - AST);
9. Patients with known retinopathy or macular degeneration;
10. Patients with history of pancreatitis;
11. Patients with concomitant use of medications that alter the absorption or excretion of azithromycin or hydroxychloroquine;
12. Breastfeeding women;
13. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of the clinical status | 15 days after randomization
  Evaluation of the clinical status of patients on the 15th day after randomization defined by the Ordinal Scale of 6 points (score ranges from 1 to 6, with 6 being the worst score)

SECONDARY OUTCOMES:
All-cause mortality | 29 days after randomization
  All-cause mortality rates at 29 days after randomization
Evaluation of the clinical status | 7 and 29 days after randomization
  Evaluation of the clinical status of patients on the 7th and 29th day after randomization defined by the Ordinal Scale of 6 points (score ranges from 1 to 6, with 6 being the worst score)
Number of days free from mechanical ventilation | 29 days after randomization
  Number of days free from mechanical ventilation at 29 days after randomization
Duration of mechanical ventilation | 29 days after randomization
  Number of days that the patient was on mechanical ventilation after randomization
Duration of hospitalization | 29 days after randomization
  Length of hospital stay on survivors
Other secondary infections | 29 days after randomization
  Presence of other secondary infections
Time from treatment start to death | 29 days after randomization
  Time from treatment start to death
Medium and long-term outcomes of SARS-CoV2 infection on morbimortality, daily life activities, mental health, and quality of life | 3, 6, 9 and 12 months
  Morbimortality, daily life activities, mental health, and quality of life
Assess whether the tested therapies may be affected by leucocyte phenotype | Baseline
  Leucocyte transcriptome

OTHER OUTCOMES:
QT interval prolongation | 29 days after randomization
  Occurrence of QT interval prolongation
Gastrointestinal intolerance | 29 days after randomization
  Occurrence of gastrointestinal intolerance
Laboratory abnormalities | 29 days after randomization
  Occurrence of laboratory hematimetric parameters, creatinine and bilirubin
Adverse events | 29 days after randomization
  Occurrence of adverse events related to the use of the investigational products

CONTACTS AND LOCATIONS:
Overall Officials: Otávio Berwanger, PhD, Study Director — Hospital Israelita Albert Einstein
Locations (58):
- Brazil (58):
  - Hospital de Urgência e Emergência de Rio Branco, Rio Branco, Acre
  - Hospital Maternidade São Vicente de Paulo, Barbalha, Ceará
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes, Fortaleza, Ceará
  - Hospital Unimed Cariri, Juazeiro do Norte, Ceará
  - Hospital Estadual Jayme dos Santos Neves, Serra, Espírito Santo
  - Hospital Evangélico de Vila Velha, Vila Velha, Espírito Santo
  - Hospital e Clínica São Roque, Ipiaú, Estado de Bahia
  - Hospital da Cidade, Salvador, Estado de Bahia
  - Hospital Brasilia, Brasília, Federal District
  - Secretaria de Estado de Saúde de Goias, Goiânia, Goiás
  - Santa Casa de Misericórdia de Belo Horizonte Santa Casa de BH, Belo Horizonte, Minas Gerais
  - Hospital Santa Paula, Passos, Minas Gerais
  - Hospital Maternidade E Pronto Socorro Santa Lucia Ltda, Poços de Caldas, Minas Gerais
  - Santa Casa da Misericordia - UTI (São João Del Rey), São João del Rei, Minas Gerais
  - Liga Paranaense de Combate ao Câncer, Curitiba, Paraná
  - Universidade Estadual de Londrina, Londrina, Paraná
  - Hospital Adventista de Belem, Belém, Pará
  - Hospital Adventista de Belém, Belém, Pará
  - Procape - Pronto S.Cardiologico de Pe.Prof.Luiz Tavares-, Recife, Pernambuco
  - Hospital Naval Marcílio Dias, Rio de Janeiro, Rio de Janeiro
  - Hospital São Lucas, Rio de Janeiro, Rio de Janeiro
  - Hospital Giselda Trigueiro, Natal, Rio Grande do Norte
  - Hospital Maternidade PROMATER, Natal, Rio Grande do Norte
  - Associação Dr. Bartholomeu Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Maestri E Kormann Consultoria Medico-Cientifica, Blumenau, Santa Catarina
  - Sociedade Literaria e Caritativa Santo Agostinho, Criciúma, Santa Catarina
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Hospital Universitário Polydoro Ernani de São Thiago/HU - UFSC, Florianópolis, Santa Catarina
  - Centro Hospitalar Unimed, Joinville, Santa Catarina
  - Hospital Dona Helena, Joinville, Santa Catarina
  - Hospital Municipal Sao Jose, Joinville, Santa Catarina
  - Hospital Regional Hans Dieter Schmidt, Joinville, Santa Catarina
  - Fundação Pio XII, Barretos, São Paulo
  - Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - nstituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Fundação do ABC (Hospital Estadual Mário Covas), Santo André, São Paulo
  - AC Camargo Cancer Center - Fundação Antonio Prudente, São Paulo, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Hospital Moriah, São Paulo, São Paulo
  - Hospital Nove de Julho, São Paulo, São Paulo
  - Hospital Santa Paula, São Paulo, São Paulo
  - Hospital São Camilo Pompeia, São Paulo, São Paulo
  - Santa Casa de Misericordia de Votuporanga, Votuporanga, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - A Beneficência Portuguesa de São Paulo - BP, São Paulo
  - Associacao Beneficente Siria, São Paulo
  - Hospital Vila Santa Catarina, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência/SP - 1, São Paulo
  - Secretaria de Saúde do Estado de São Paulo, São Paulo
  - Serv Social da Industria do papel, papelão e cortiça do estado de SP, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sírio-Libanês, São Paulo
  - Universidade Federal de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furtado RHM, Barros E Silva PGM, Fonseca HAR, Serpa-Neto A, Correa TD, Guimaraes HP, Pereira AJ, Olivato GB, Zampieri FG, Lisboa T, Junqueira DLM, Lapa MG, Monfardini F, Damiani LP, Echenique LS, Gebara OE, Hoffman Filho CR, Polanczyk CA, Rohde LE, Amazonas R, Machado FR, Avezum A, Azevedo LCP, Veiga VC, Rosa RG, Lopes RD, Cavalcanti AB, Berwanger O; COALITION COVID-19 Brazil Steering Committee and Investigators. Cardiovascular Safety of Azithromycin in Patients Hospitalized With COVID-19: A Prespecified Pooled Analysis of the COALITION I and COALITION II Randomized Clinical Trials. Am J Cardiol. 2024 Mar 1;214:18-24. doi: 10.1016/j.amjcard.2023.11.069. Epub 2023 Dec 15. PMID 38104755
- [Derived] Furtado RHM, Berwanger O, Fonseca HA, Correa TD, Ferraz LR, Lapa MG, Zampieri FG, Veiga VC, Azevedo LCP, Rosa RG, Lopes RD, Avezum A, Manoel ALO, Piza FMT, Martins PA, Lisboa TC, Pereira AJ, Olivato GB, Dantas VCS, Milan EP, Gebara OCE, Amazonas RB, Oliveira MB, Soares RVP, Moia DDF, Piano LPA, Castilho K, Momesso RGRAP, Schettino GPP, Rizzo LV, Neto AS, Machado FR, Cavalcanti AB; COALITION COVID-19 Brazil II Investigators. Azithromycin in addition to standard of care versus standard of care alone in the treatment of patients admitted to the hospital with severe COVID-19 in Brazil (COALITION II): a randomised clinical trial. Lancet. 2020 Oct 3;396(10256):959-967. doi: 10.1016/S0140-6736(20)31862-6. Epub 2020 Sep 5. PMID 32896292
- [Derived] Lasheras I, Santabarbara J. Use of antimalarial drugs in the treatment of COVID-19: A window of opportunity? Med Clin (Barc). 2020 Jul 10;155(1):23-25. doi: 10.1016/j.medcli.2020.04.004. Epub 2020 Apr 22. No abstract available. English, Spanish. PMID 32386744